CLINICAL TRIAL: NCT03492710
Title: Phase III Study of Immune Globulin Intravenous (Human) IGIV-SN in Pediatric Subjects With Primary Humoral Immunodeficiency
Brief Title: Study of Immune Globulin Intravenous (Human) GC5101F in Subjects With Primary Humoral Immunodeficiency
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: A change in sponsor's developmental strategy
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC5101F
Record Dates: First submitted 2018-02-19; First posted 2018-04-10 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Primary Immune Deficiency Disorder
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Immunoglobulins

STUDY DESIGN:
Intervention Model Description: Open-Label, Single-Arm, Historically Controlled, Prospective, Multicenter
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IGIV-SN (Experimental): Immunoglobulin, Supplied in 5g (100mL) and/or 10g (200mL)
  Interventions: Biological: Immunoglobulin

INTERVENTIONS:
Biological: Immunoglobulin — Administer volume of IGIV-SN to maintain a trough level of of 5g/L or more
  Other Names: IGIV-SN

SUMMARY:
To assess the safety, efficacy, and pharmacokinetics of IGIV-SN in pediatric subjects with primary immunodeficiency humoral diseases (PHID)

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects with a confirmed clinical diagnosis of a Primary Humoral Immunodeficiency Disease as defined by IUIS (International Union of Immunological Societies) and require treatment with IGIV. Documented agammaglobulinemia or hypogammaglobulinemia
* Subject is willing to comply with all requirements of protocol
* Authorization to access personal health information

Exclusion Criteria:

* Subject has secondary immunodeficiency
* Subject has a history of repeated reactions or hypersensitivity to IGIV or other injectable forms of IgG
* Subject has significant protein loss from enteropathy, nephrotic syndrome or lymphangiectasia

Ages: 24 Months to 203 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy: Incidence of Acute SBIs (Serious Bacterial Infections) | 13 months (12 months of treatment + 1 month of Follow-Up)
  The incidence of acute serious bacterial infections, i.e. bacterial pneumonia, bacteremia/sepsis, bacterial meningitis, osteomyelitis/ septic arthritis, visceral abscess
Safety: Overall Incidence of AEs that occur during 72 hours of following an infusion of test drug | 13 months (12 months of treatment + 1 month of Follow-Up)
  The overall incidence of adverse events (AEs) that occur during or within 1 hours, 24 hours, and 72 hours following an infusion of test product, regardless of whether or not the AE is determined to be product related

SECONDARY OUTCOMES:
Efficacy: Incidence of Infections other than acute serious bacterial infections | 13 months (12 months of treatment + 1 month of Follow-Up)
Safety: The frequency of all AEs that occuring during the study | 13 months (12 months of treatment + 1 month of Follow-Up)
  (regardless of the casual relationship)

OTHER OUTCOMES:
PK Endpoint (1) | 13 months (12 months of treatment + 1 month of Follow-Up)
  Plasma Concentration-Time Curve (PK Parameters of Total IgG)
PK Endpoint (2) | 13 months (12 months of treatment + 1 month of Follow-Up)
  Area Under the Curve (PK Parameters of Total IgG)

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Roifman, Principal Investigator — The Hospital for Sick Children